CLINICAL TRIAL: NCT04486534
Title: The Assessment of Talar Cartilage, Tibialis Antetior and Gastrocnemius Muscles in Patients With Unilateral Traumatic Transtibial Amputation: a Clinical and Sonographic-controlled Study
Brief Title: The Assessment of Talar Cartilage in Patients With Unilateral Traumatic Transtibial Amputation
Status: Completed | Type: Observational
Sponsor: Gaziler Physical Medicine and Rehabilitation Education and Research Hospital (Other)
Responsible Party: Principal Investigator, Yasin Demir, Physical Medicine and Rehabilitation Specialist, Gaziler Physical Medicine and Rehabilitation Education and Research Hospital
Other Study IDs: 4
Record Dates: First submitted 2020-07-16; First posted 2020-07-24 (Actual); Last update posted 2021-02-17 (Actual); Status verified 2021-02

CONDITIONS: Traumatic Amputation of Lower Extremity; Cartilage Degeneration
Keywords: Amputation; Transtibial; Prosthesis; Cartilage; Muscle

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Case group: 36 patients between the ages of 18-65, who have been followed up for at least 3 months with the diagnosis of unilateral transtibial amputation and who have been using prostheses for at least 3 months
  Interventions: Other: Musculoskeletal ultrasound
- Control group: 36 age and body mass index (BMI)-matched healthy controls
  Interventions: Other: Musculoskeletal ultrasound

INTERVENTIONS:
Other: Musculoskeletal ultrasound — Subjects' talar cartilage, tibialis anterior and gastrocnemius muscle thickness measurements will be performed using musculoskeletal ultrasound.

SUMMARY:
Increased risk of osteoarthritis (OA) has been previously demonstrated in patients with lower limb amputation. Although there are many studies on knee joint of intact limb of amputees in the literature, the number of studies on intact foot and ankle is extremely limited. The primary aim of the study is to compare the intact talar cartilage, tibialis anterior and gastrocnemius muscle thickness measurements of traumatic unilateral transtibial amputee patients with that of healthy individuals using ultrasound. The secondary aim is to investigate the relationship between cartilage and muscle thickness measurements with clinical parameters.

DETAILED DESCRIPTION:
Methods: A total of 36 patients with unilateral transtibial amputations and 36 age and body mass index (BMI)-matched male controls will be participated in this cross-sectional study. Functional performance will be assessed by 6-minute walking distance (in meter). The Foot and Ankle Outcome Score (FAOS) will be used for the assessment of the symptoms and the functional limitations of the foot and ankle. The health-related quality of life of the subjects will be evaluated with Short Form-36 (SF-36). Subjects' talar cartilage, tibialis anterior and gastrocnemius muscle thickness measurements will be performed using musculoskeletal ultrasound.

ELIGIBILITY:
Inclusion Criteria:

* Patients between the ages of 18-65
* Patients who have been followed up for at least 3 months with the diagnosis of unilateral transtibial amputation
* Patients who have been using prostheses for at least 3 months

Exclusion Criteria:

* Bilateral amputation
* Previous history of any trauma/surgical history of the lower extremities (other than amputation)
* Rheumatic diseases
* Contracture of the knee and the ankle of the intact limb

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: A total of 36 patients with unilateral transtibial amputations and 36 age and BMI-matched healthy controls
Sampling Method: Non-Probability Sample
Enrollment: 72 (Actual)
Dates: Start 2020-07-26 (Actual); Primary Completion 2021-01-15 (Actual); Study Completion 2021-01-15 (Actual)

PRIMARY OUTCOMES:
Talar cartilage, tibialis anterior and gastrocnemius muscle thickness measurements | through study completion, an average of one and a half months
  Talar cartilage, tibialis anterior and gastrocnemius muscle thickness measurements will be performed by using ultrasound.

SECONDARY OUTCOMES:
6-minute walking test | through study completion, an average of one and a half months
  Functional performance will be assessed by 6-minute walking distance (in meter)
The Foot and Ankle Outcome Score (FAOS) | through study completion, an average of one and a half months
  The Foot and Ankle Outcome Score (FAOS) will be used for the assessment of the symptoms and the functional limitations of the foot and ankle. The FAOS consists of 42 questions, divided into five different patient-relevant subscales: pain (nine questions); symptoms such as stiffness, swelling and range of motion (seven questions); activities of daily living (17 questions); ability to perform sports and recreational activities (five questions); and foot/ankle-related quality of life (four questions). Answers are given on a five-point Likert scale. Total and subscores are calculated by summing the scores of the individual items. The total score is recoded into a 0-100 scale, with 100 representing no symptoms or limitations.
Short Form-36 (SF-36) | through study completion, an average of one and a half months
  The health-related quality of life of the subjects will be evaluated with Short Form-36 (SF-36). This comprises 36 questions related to eight different subscales, physical functioning, bodily pain, role limitation, due to physical health problems, general health perceptions, vitality, energy and fatigue, role limitations due to emotional problems, social functioning and general mental health, which covers psychological distress and wellbeing. Each of eight subscales is scored between 0 and 100, with higher scores indicating a better quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Merve Orucu Atar, MD, Principal Investigator — Gaziler PMR, Training and Research Hospital, Department of PMR
Locations (1):
- Merve Orucu Atar, Ankara, Cankaya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Orucu Atar M, Bilgin E, Demir Y, Korkmaz N, Gurcay E. Comparison of thicknesses of talar cartilage, tibialis anterior, and gastrocnemius muscles between high-activity patients with unilateral traumatic transtibial amputation and nonamputated individuals: A clinical and sonographic study. Prosthet Orthot Int. 2022 Oct 1;46(5):459-465. doi: 10.1097/PXR.0000000000000159. Epub 2022 Jul 1. PMID 36215056